CLINICAL TRIAL: NCT03169309
Title: The BEST Study: The Efficacy of Brain Entrainment Sleep Technology in Military Healthcare Beneficiaries
Acronym: BEST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study modified to a two-group crossover design and transferred to new location.
Sponsor: Landstuhl Regional Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr MeLisa Gantt, (former) Chief, CNSCI, Landstuhl Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: M-10544
Record Dates: First submitted 2017-03-07; First posted 2017-05-30 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Sleep; Sleep Disorders; Sleep Deprivation; Sleep Disturbance; Sleep Disorders, Intrinsic; Sleep Disorders, Circadian Rhythm
Keywords: complementary and alternative medicine; military; binaural beat technology; brain entrainment technology; sleep
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Deprivation; Parasomnias; Sleep Disorders, Intrinsic; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: Pre- and post- intervention trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre and Post Intervention (Experimental): One Study Arm - Quantitative and qualitative sleep quality measure will be captured at baseline (Phase I/Week 1-2), while using Brain Entrainment Technology (Phase II/Week3-4), and after using the technology.
  Interventions: Device: Brain Entrainment Technology

INTERVENTIONS:
Device: Brain Entrainment Technology — Brain Entrainment Technology (BET), also known as Binaural Beat Technology (BBT), is a sound technology where two slightly different tones are present to each ear and the brain produces a third tone. This third tone impacts the reticular activating system which alters the action potentials of the thalamus and cerebral cortex in turn changing the brain wave frequency to alter the state of consciousness of the listener.
  Other Names: Binaural Beat Technology

SUMMARY:
Brain Entrainment Technology (BET), also known as Binaural Beat Technology (BBT); is an auditory-neurophysiologic technique which uses auditory tones (often embedded in music, nature sounds or white noise) dichotically via stereo headphones to manipulate brainwave activity in turn affecting the listener's mental, physical and/or emotional state. Although this technology is widely marketed to the general public and can be found free in on the internet, only a hand full of scientific studies have shown its efficacy. This study is a follow-on study to the "Sound Mind Warrior (SMW) Study" (ClinicalTrials.gov [NCT02328690]) conducted 2012-2015 which assessed the efficacy of the technology (in the "theta" brainwave frequency) on the cardiovascular stress response in a group of service members with complaint of chronic stress. This study will now assess BET (in the "delta" brainwave frequency) on sleep quality in a population of military healthcare beneficiaries with complaint of poor sleep quality.

DETAILED DESCRIPTION:
This study will follow a prospective, one group pre- and post-intervention design.

A sample of 162 military healthcare beneficiaries (within the Kaiserslautern Military Community footprint) with complaints of poor sleep quality will be instructed to wear sleep actigraphy monitors and complete daily sleep diaries upon waking for a total of four weeks. On weeks 3 and 4, participants will use BET at bedtime for a minimum of 30 minutes. Pre and post sleep quality measures will be compared along with pre- and post- c-reactive protein (CRP) measures and a post-study questionnaire to assess participants' perception about the technology.

ELIGIBILITY:
Inclusion Criteria:

* Score greater than or equal to 15 on the Insomnia Severity Index (ISI)
* Affiliated with at least one of the 13 installations within the Kaiserslautern Military Community (KMC) area
* Eligible to receive healthcare at Landstuhl Regional Medical Center (LRMC)
* Are 18 years or older
* Can read and speak English
* Are able to commit to a 4 week study

Exclusion Criteria:

* Are taking any type of medication that causes drowsiness
* Have been diagnosed with moderate to severe traumatic brain injury (TBI)
* Have a history of epilepsy
* Are taking any medication in the anti-seizure category
* Have been diagnosed with, taking medication for, or are currently being evaluated for a psychological health issue as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) that will prohibit them from using intervention as perscribed.
* Have ear trauma, difficulty hearing or wear a hearing aide
* Have a chronic inflammatory health issue
* Are pregnant or are trying to become pregnant in the next 4 weeks

  *Women of child bearing age will be asked to provide a urine sample for a pregnancy test
* Are currently using BET

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
"Quantitative" Sleep Quality (via Sleep Actigraphy Watch) | Daily over the course of 4 weeks
  Sleep actigraphy monitor will measure wake/sleep. Using special software, that information is then articulated into graphical and tabulated report that shows the movement that occurred throughout the wake and sleep cycles as well as light exposure that may have affected sleep. The report gives the a) time the participants went to bed, b) time they woke up, c) number of hours they were in the bed, d) total number of hours asleep, e) number of minutes it took to fall asleep, f) percent efficiency of their sleep, g) number of minutes awaken after sleep onset, and h) total number of times they woke up after falling asleep.

SECONDARY OUTCOMES:
Insomnia Severity Level (via Insomnia Severity Index Questionnaire) | Baseline
  A 7-item questionnaire will be used as a screening tool to quantify the severity level of the participant's poor sleep quality. It is comprised of a 5-point Likert scale with a total score from 0-28 with 15 or greater indicating moderate to severe insomnia
"Qualitative" Sleep Quality (via Sleep Foundation Sleep Diary Questionnaire) | Daily over the course of 4 weeks
  A 14-item questionnaire will be used to capture sleep habits. Questions cover: napping, caffeine, alcohol, exercise, medication, meals, sleepiness, sleep hygiene, and quality. This instrument is not scored but merely used to assess patterns and if those patterns changed over the course of the study.
Overall Impression of Sleep Quality (via Pittsburgh Sleep Quality Index Questionnaire) | Baseline and Week 4 (after using intervention)
  A 24-item item questionnaire gives an accumulative score based on sub scores of sleep duration, sleep disturbance, sleep latency, number of days of dysfunction due to sleepiness, sleep efficiency, sleep quality, and medication usage. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: TOTAL < 5 associated with good sleep quality and TOTAL > 5 associated with poor sleep,
Inflammatory Biomarker (via C-Reactive Protein Lab) | Baseline and Week 4 (after using intervention)
  A blood sample for c-reactive protein will measures the inflammatory process. After accounting for any external influences on CRP level, this measure will be correlated with the objective and subjective sleep data to assess if changes in sleep quality affected the inflammatory response.
Extenuating Factor Affecting C-Reactive Protein Level (via C-Reactive Protein Questionnaire) | Baseline and Week 4 (after using intervention)
  Since exposure to stress, infection, allergy, injury, or menstruation could affect CRP levels; this 6-item questionnaire will be used to note other possible co-variates that could have impacted CRP levels.
Overall Impression of Brain Entrainment Technology (via Post Study Questionnaire) | Week 4 (after using intervention)
  A 10-item questionnaire will be used at the completion of the study to instrument will capture any subjective comments from the participants as to assess the participant's perception about the technology as well as to assess ways that will help improve future studies using the same equipment and/or technology.

CONTACTS AND LOCATIONS:
Overall Officials: MeLisa Gantt, PhD, Principal Investigator — Gantt Clinical Institute LLC
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Germany

IPD SHARING:
Plan to Share IPD: No